CLINICAL TRIAL: NCT01407965
Title: Offene, Monozentrische, Nicht Kontrollierte Und Nicht Randomisierte Phase IV-Studie Zur Bestimmung Der Pharmakokinetik Von Carbapenemen in adipösen Patienten.
Brief Title: Pharmacokinetics of Carbapenem Antibiotics in Obese Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, M. Wittau, MD, University of Ulm
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Adip-2010; 2010-024094-39 (EudraCT Number)
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: obesity; pharmacokinetic; ertapenem; meropenem
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ertapenem (Experimental): Free tissue kinetics of ertapenem in fatty tissue and intraperitoneal fluid in mg/L
  Free and bound plasma concentration of ertapenem or meropenem in mg/L
  Interventions: Procedure: microdialysis catheter
- Meropenem (Experimental): Free tissue kinetics of meropenem in fatty tissue and intraperitoneal fluid in mg/L up to 24 hours after administration. Free and bound plasma concentration of meropenem in mg/L.
  Interventions: Procedure: microdialysis catheter

INTERVENTIONS:
Procedure: microdialysis catheter — Placing of microdialysis catheter in fatty tissue and in the peritoneal cavity
  Arms: Ertapenem
Procedure: microdialysis catheter — Placing of microdialysis catheter in fatty tissue and in the peritoneal cavity
  Arms: Meropenem

SUMMARY:
Tissue kinetics of ertapenem and meropenem in fatty tissue, intraperitoneal fluid and plasma.

DETAILED DESCRIPTION:
The purpose of this study is to determine the free tissue kinetics of ertapenem and meropenem in fatty tissue and intraperitoneal fluid up to 24 hours after administration of the IMP.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients 18 years or older requiring elective surgical intervention (open or laparoscopic surgery) at intraabdominal organs
* BMI more or even 40
* written informed consent

Exclusion Criteria:

* BMI < 40
* pregnancy or lactation in women
* emergency surgery
* history of serious allergy or intolerance to β-lactam antibiotics
* systemic antimicrobial therapy with ceftazidime (internal standard of high-performance liquid chromatography / mass spectrometry) within a 7 days period prior to study entry
* ongoing intraabdominal infections
* terminal illness
* severe diseases of the liver, e.g. cirrhosis of the liver with ALT or AST > 6 x upper limit of normal (ULN) and bilirubin > 3 x ULN
* severe renal insufficiency with a creatinine clearance ≤30 mL/min.
* neutrophil count < 1000 cells/mm3
* platelets < 75000 cells/mm3
* coagulation studies (INR) > 1.5 x ULN
* ongoing chemotherapy and/or radiotherapy
* ongoing therapy with valproin acid (in case of ertapenem administration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Unbound concentration of ertapenem and meropenem in fatty tissue and peritoneal fluid | within 24 h after administration

SECONDARY OUTCOMES:
Number of Adverse Events (total and per patient) | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Number of Serious Adverse Events (total and per patient) | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Number of Suspected Unexpected Serious Adverse Reactions (SUSARs) | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doris Henne-Bruns, PhD, Principal Investigator — University of Ulm; Mathias Wittau, Dr., Principal Investigator — University of Ulm
Locations (2):
- Germany (2):
  - University of Ulm, Dept. of Visceral Surgery, Ulm
  - University of Ulm, Ulm

REFERENCES:
- [Derived] Wittau M, Paschke S, Kurlbaum M, Scheele J, Ly NS, Hemper E, Kornmann M, Henne-Bruns D, Bulitta JB. Population Pharmacokinetics and Target Attainment of Ertapenem in Plasma and Tissue Assessed via Microdialysis in Morbidly Obese Patients after Laparoscopic Visceral Surgery. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e00952-16. doi: 10.1128/AAC.00952-16. Print 2017 Jan. PMID 27795367
- [Derived] Wittau M, Scheele J, Kurlbaum M, Brockschmidt C, Wolf AM, Hemper E, Henne-Bruns D, Bulitta JB. Population Pharmacokinetics and Target Attainment of Meropenem in Plasma and Tissue of Morbidly Obese Patients after Laparoscopic Intraperitoneal Surgery. Antimicrob Agents Chemother. 2015 Oct;59(10):6241-7. doi: 10.1128/AAC.00259-15. Epub 2015 Jul 27. PMID 26248353